CLINICAL TRIAL: NCT00847769
Title: Effect of Manual Therapy Intervention on Corticospinal Excitability in Individuals With Post-acute Ankle Sprains
Brief Title: Ankle Sprains and Corticospinal Excitability
Acronym: ACE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of the Pacific (Other); American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Beth Fisher, Co-Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HS-08-00192
Record Dates: First submitted 2009-01-22; First posted 2009-02-19 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Ankle Sprain
Keywords: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Traction; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High velocity, low amplitude stretch (Experimental): With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. A thrust will be delivered parallel to the long axis of the subject's lower leg after the treating therapist induces passive ankle dorsiflexion to end range.
  Interventions: Other: High velocity, low amplitude stretch
- Slow, mobilization stretch (Active Comparator): With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. Traction will be delivered to the talocrural joint at the treating therapist's second perception of tissue resistance in 3 bouts of 30-second holds, separated by 10 seconds of rest.
  Interventions: Other: Slow, mobilization stretch
- Passive positioning (Sham Comparator): With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface, which is similar to the positioning used for the active comparator groups. The treating investigator will maintain passive positioning of the ankle for the duration of 1 deep inhalation and exhalation by the subject rather than induce an iatrogenic force.
  Interventions: Other: Passive Positioning

INTERVENTIONS:
Other: High velocity, low amplitude stretch — This group (n=9) will receive talocrural traction manipulation. With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. A thrust will be delivered parallel to the long axis of the subject's lower leg after the treating therapist induces passive ankle dorsiflexion to end range.
  Other Names: Manipulation; GPM-V
  Arms: High velocity, low amplitude stretch
Other: Slow, mobilization stretch — This group (n=9) will receive talocrural traction mobilization. With the subject in a seated position on a treatment table and the lower extremity of interest stabilized to the table with a belt, a single standardized treating investigator will grasp the foot of interested with the thenar eminences on the foot's plantar surface. Traction will be delivered to the talocrural joint at the treating investigator's second perception of tissue resistance in 3 bouts of 30-second holds, separated by 10 seconds of rest.
  Other Names: Articulation; Mobilization; Traction
  Arms: Slow, mobilization stretch
Other: Passive Positioning — This group (n=9) will receive the manual therapy control intervention. This will consist of the same patient and clinician preparation for the mobilization/manipulation techniques. However, a single standardized treating investigator will simply maintain passive ankle positioning for the duration of 1 deep inhalation and exhalation by the subject rather than induce an iatrogenic force characteristic of the intervention received by the other 2 comparison groups.
  Other Names: Passive Range of Motion; Placebo
  Arms: Passive positioning

SUMMARY:
The purpose of this study is to determine changes in the brain associated with improvement in ankle range of motion following ankle manual therapy procedures in individuals with post-acute ankle sprains

DETAILED DESCRIPTION:
Physical therapists use many ways to treat joints that do not move well. One way takes 1-2 seconds. Another way may take up to 1 minute. Both stretches seem to work, but we do not know how. Certain changes in the brain and spinal cord may cause joints to become more flexible after these kinds of stretches. Right now, we do not have very much information about how these might work in people who have injured their ankle. This study will find out if changes in the brain cause better flexibility in the ankle joint after different kinds of stretches. In this study, subjects with a certain kind of ankle sprains and limited ankle joint flexibility will be assigned to 1 out of 3 groups. Subjects will not get to choose their groups. The first group will have an ankle stretch that lasts 1-2 seconds. The second group will have a stretch that last 1 minute. The third group will have their foot held without any stretching. We will use a machine to stimulate the brain and spinal cord to find out how these stretches affect the brain and spinal cord. The machine sends a magnetic signal to the brain, and we will measure how much signal gets through to the leg muscles using electrodes on the skin. We also will use 3 flexibility tests to find out how well each stretch worked. One test is with the subject lying on their stomach, and the others are with the subject standing up. To start the study, subjects will get their brain stimulated. They will then get their brain stimulated again one hour later. After the second stimulation, subjects will have their flexibility tested and then get 1 of the 3 treatments. After the treatment, subjects will get a last brain stimulation test and flexibility tests. We think subjects that get a fast stretch will have better brain function and flexibility than subjects that get the slow stretch or no stretch. To test our idea, we will compare how each group did with the brain stimulation and flexibility tests. We will also look at the relationship between brain function and flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Onset of ankle sprain at least 2 weeks prior to enrollment
* Foot and Ankle Ability Measure Activity of Daily Living subscale score less than or equal to 80%
* Ankle dorsiflexion range of motion less than or equal to 5 degrees

Exclusion Criteria:

* Current status of assisted ambulation (eg, use of cane or crutches)
* Inability to bear weight through the affected extremity immediately after injury combined with tenderness to palpation of the medial and lateral malleolar zones, styloid process of the 5th metatarsal, and navicular
* Positive anterior drawer or talar tilt dimple test
* Volume of the affected limb greater than 10% of the unaffected limb
* Previous history of ligament or bony reconstructive surgery to the ankle and foot
* Concomitant injury to other lower extremity joints
* Medical conditions that serve as contraindications to mobilization/manipulation and transcranial magnetic stimulation, such as presence of pacemaker, metal in head, pregnancy, neurological disorders, recent use of stimulants or medications known to lower seizure threshold, and personal or family history of seizures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Corticospinal motor excitability (transcranial magnetic stimulation variables) | Pre-intervention measurement, 1 additional repeated pre-intervention measurement, post-intervention measurement

SECONDARY OUTCOMES:
Single leg squat reach test | Pre-intervention measurement, 1 additional repeated pre-intervention measurement, post-intervention measurement
Ankle flexibility test (laying on stomach) | Pre-intervention measurement, 1 additional repeated pre-intervention measurement, post-intervention measurement
Ankle flexibility test (standing against wall) | Pre-intervention measurement, 1 additional repeated pre-intervention measurement, post-intervention measurement

CONTACTS AND LOCATIONS:
Overall Officials: Beth E Fisher, PhD, PT, Principal Investigator — University of Southern California; Todd E Davenport, DPT, OCS, Study Director — University of the Pacific
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Fisher BE, Piraino A, Lee YY, Smith JA, Johnson S, Davenport TE, Kulig K. The Effect of Velocity of Joint Mobilization on Corticospinal Excitability in Individuals With a History of Ankle Sprain. J Orthop Sports Phys Ther. 2016 Jul;46(7):562-70. doi: 10.2519/jospt.2016.6602. Epub 2016 Jun 6. PMID 27266885
- [Derived] Fisher BE, Davenport TE, Kulig K, Wu AD. Identification of potential neuromotor mechanisms of manual therapy in patients with musculoskeletal disablement: rationale and description of a clinical trial. BMC Neurol. 2009 May 21;9:20. doi: 10.1186/1471-2377-9-20. PMID 19460169